CLINICAL TRIAL: NCT04820322
Title: Comparison of Postprandial Glycemic and Insulinemic Response to a Cookie With or Without Added Fibersym After Three Days of Pre-feeding: An Acute Double-blind, Randomized Controlled Clinical Trial
Brief Title: Comparison of the Postprandial Glycemic and Insulinemic Response After a Fibersym Containing Cookie With a Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MGP Ingredients, Inc. (Industry)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Principal Investigator, Dr. Thomas M. Wolever, President, Glycemic Index Laboratories, Inc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: GIL-1852
Record Dates: First submitted 2021-02-23; First posted 2021-03-29 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Postprandial Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Intervention Model Description: double blind, controlled, cross-over clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The product was re-packaged by a GI Labs staff member not involved in the clinical trial. Product label displayed the subject number, subject initials, product ID, ingredients statement, GIL repacked date, expiration date, researcher name and telephone number, investigational use statement, and allergy warnings. After the data had been entered, checked for errors and the database locked, the code was broken, #149 corresponded to the control cookie while 394 corresponded to the Fibersym cookie..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control cookie (Placebo Comparator): a sugarsnap cookie baked specifically for this trial
  Interventions: Other: Control cookie
- Fibersym cookie (Active Comparator): a sugarsnap cookie baked using the same methodology for the control cookie but with the resistants starch RS4, Fibersym, added
  Interventions: Other: Fibersym

INTERVENTIONS:
Other: Fibersym — RS4-type resistant modified wheat starch
  Arms: Fibersym cookie
Other: Control cookie — control cookie
  Arms: control cookie

SUMMARY:
Fibersym® is a RS4-type resistant modified wheat starch in which over 85% of the total starch is resistant starch as measured by AOAC method 991.43. It is meant to be consumed on a regular basis and doses up to 33g/day can be tolerated. The effect of a Fibersym-containing meal on postprandial glucose and insulin levels when compared to a control meal, where both meals contain the same amount of available carbohydrate, is not known. This study therefore investigated the acute effect of a Fibersym cookie and a control cookie matched for available carbohydrate after a 3-day habituation period.

DETAILED DESCRIPTION:
The study used a double-blind, randomized, cross-over design.

Visit 1: Participants willing to be considered were invited to come to the research centre to have the study procedures explained to them and be given a copy of the consent form which they may either sign then, take away to sign at a later date, or decline to participate. Participants were encouraged to ask any questions they may have and not to sign the consent form until all of their questions have been answered to their satisfaction. Those who consented to participate came to the research centre for a pre-selection visit when subject eligibility will be determined. A number of parameters were assessed including blood pressure, weight, height, BMI, and brief medical history.

Visit 2-3: Each eligible subject received one of the treatments at visit 2 and the other at visit 3. The order of the 2 treatments was randomized using an online randomization calculator. The interval between visits was no less than 6 days and no more than 4 weeks. Prior to each visit there was a 3-day pre-feeding period during which subjects consumed either 108.9g Control Cookies (approx. 3.5 cookies) per day or 136.2 g of Fibersym Cookies (approx. 4 cookies) per day (delivering 29 g fiber from Fibersym/day) according to the randomized order. Cookies were consumed with each main meal (breakfast, lunch and dinner).

Subjects were provided with a calorie appropriate, standard frozen dinner to be consumed on the evening before each visit. On the day of each visit, participants came to GI Labs in the morning after a 10-12 h overnight fast (except for water). Two (2) fasting fingerprick blood samples were collected at -5 min and 0 min. Each sample consisted of 2 vials, one for glucose analysis and one for insulin analysis (4-8 drops of blood each). Questionnaires to record satiety and GI symptoms were administered. Participants were then a 40g available carbohydrate protion of the same type of cookie (Control or Fibersym) they had been consuming over the past 3 days containing together with 250 ml of water and instructed to consume them over 15 minutes. Additional blood samples were collected 15, 30, 45, 60, 90 and 120 min after the start of the test meal. Satiety questionnaires were administered at the same time intervals. GI symptom questionnaires were filled out at 2 h in addition to fasting.

Test Foods:

The sugar snap cookie formula (Control) was obtained from the American Institute of Baking (AIB) International (Manhattan, KS). Fibersym RW (Appendix 1) was added as an extra portion to the Control Cookie recipe, amounts were adjusted so that both the control and Fibersym cookie portions contained the same amount of available carbohydrate (ingredients are listed in appendix 1). Both cookies were baked at the facilities of AIB. The macronutrient composition of baked cookies was determined by an independent laboratory and the final weights of the cookies fed were adjusted accordingly.

To maintain blinding, the cookies were re-packaged by a GI Labs staff member not involved in the clinical trial. Product label displayed the subject number, subject initials, product ID, ingredients statement, GIL repacked date, expiration date, researcher name and telephone number, investigational use statement, and allergy warnings (if needed). Study Product Intake Logs were completed upon dispensation of study product to each subject. After the data had been entered, checked for errors and the database locked, the code was broken.

Participants were asked to maintain stable dietary and activity habits throughout their participation and to refrain from drinking alcohol and from unusual levels of food intake or physical activity for 24 h before each test. Subjects were asked to complete a 3- day record of supplement consumption and whether they consumed the standard evening meal, in addition to a 3-day symptom diary before each test visit. If any subject was not feeling well or had not complied with the preceding experimental conditions, the test was not carried out and was rescheduled for another day.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant females, 18-75 years of age, inclusive
* Body mass index (BMI) between 18.5 and 35 kg/m² inclusive at screening.
* Systolic blood pressure <130 mm Hg; Diastolic blood pressure <90 mm Hg.
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
* Willing to abstain from strenuous exercise, or consume alcoholic drinks 24 hours before study days.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study Investigator.
* Female subjects; willing to use a contraceptive method to avoid pregnancy during the study period.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Smokers
* Known history of diabetes, gastrointestinal, liver, kidney, or cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), and pulmonary disease
* Use of medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might, in the opinion of Dr. Wolever, the president of GI Testing, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Use of antibiotics within 4 weeks of start of study
* Major trauma or surgical event within 3 months of screening.
* Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
* Known intolerance, sensitivity or allergy to any ingredients in the study products.
* Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.)
* Change in body weight of >3.5 kg within 4 weeks of the screening visit.
* History of cancer in the prior two years, except for non-melanoma skin cancer.
* Exposure to any non-registered drug product within 30 d prior to screening.
* Pregnancy or breastfeeding
* Any history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, binge eating) diagnosed by a health professional

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wolever TMS, Maningat CC, Seib PA, Campbell JE, Jenkins AL. Cross-linked phosphorylated RS4 wheat starch reduces glucose and insulin responses after 3 days of pre-feeding in healthy adults: an acute, double-blind, randomized controlled clinical trial. Int J Food Sci Nutr. 2023 Sep;74(5):621-629. doi: 10.1080/09637486.2023.2236809. Epub 2023 Jul 20. PMID 37475127

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized to the treatment order on the first visit after screening. None were excluded between screening and the first visit. Ten (n=10) participants were randomized to receive the control cookie first followed by the Fibersym cookie; one participant dropped out after the control cookie due to developing and infection. Six (n=6) participants were randomized to receive the fibersym cookie first followed by the control cookie.
Groups:
- Experimental: Control Cookie, Then Fibersym Cookie: Participants consumed 109g of control cookies (about 3.5 cookies - at least 1 cookie at each main meal) daily for 3 days. On the evening of the 3rd day they consumed the frozen dinner they had been provided with. They came to the test center the next morning after an overnight fast when the glucose and insulin responses elicited by 78.1g of control cookie (40g available carbohydrate) were measured. After a 6-28 day washout period participants repeated the process, consuming 136g of Fibersym cookies (about 4 cookies, 29g fiber, at least 1 with each main meal) daily for 3 days, consuming the standard dinner on the 3rd day and after an overnight fasting having glucose and insulin responses elicited by 97.8g Fibersym cookie (40g available carbohydrate) measured.
- Fibersym Cookie First: Participants consumed 136g of Fibersym cookies (about 4 cookies, 29g fiber, at least 1 cookie at each main meal) daily for 3 days. On the evening of the 3rd day they consumed the frozen dinner they had been provided with. They came to the test center the next morning after an overnight fast when the glucose and insulin responses elicited by 97.8g of Fibersym cookie (40g available carbohydrate) were measured. After a 6-28 day washout period participants repeated the process, consuming 109g of control cookies (about 3.5 cookies, at least 1 with each main meal) daily for 3 days, consuming the standard dinner on the 3rd day and after an overnight fasting having glucose and insulin responses elicited by 78.1g Control cookie (40g available carbohydrate) measured.
Period: Overall Study
Arm/Group | Experimental: Control Cookie, Then Fibersym Cookie | Fibersym Cookie First
Started | 10 | 6
Completed | 9 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: 15 completed the cross-over study successfully and all were included in the analysis
Groups:
- Control Cookie First Followed by Fibersym Cookie: Participants consumed 109g of control cookies (about 3.5 cookies - at least 1 cookie at each main meal) daily for 3 days. On the evening of the 3rd day they consumed the frozen dinner they had been provided with. They came to the test center the next morning after an overnight fast when the glucose and insulin responses elicited by 78.1g of control cookie (40g available carbohydrate) were measured. After a 6-28 day washout period participants repeated the process, consuming 136g of Fibersym cookies (about 4 cookies, 29g fiber, at least 1 with each main meal) daily for 3 days, consuming the standard dinner on the 3rd day and after an overnight fasting having glucose and insulin responses elicited by 97.8g Fibersym cookie (40g available carbohydrate) measured.
- Fibersym Cookie First Followed by Control Cookie: Participants consumed 136g of Fibersym cookies (about 4 cookies, 29g fiber, at least 1 cookie at each main meal) daily for 3 days. On the evening of the 3rd day they consumed the frozen dinner they had been provided with. They came to the test center the next morning after an overnight fast when the glucose and insulin responses elicited by 97.8g of Fibersym cookie (40g available carbohydrate) were measured. After a 6-28 day washout period participants repeated the process, consuming 109g of control cookies (about 3.5 cookies, at least 1 with each main meal) daily for 3 days, consuming the standard dinner on the 3rd day and after an overnight fasting having glucose and insulin responses elicited by 78.1g Control cookie (40g available carbohydrate) measured.
- Total: Total of all reporting groups
Arm/Group | Control Cookie First Followed by Fibersym Cookie | Fibersym Cookie First Followed by Control Cookie | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (12) | 29 (8) | 31 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: 2-hour Postprandial Glucose Incremental Area Under the Curve (IAUC)
Description: 2-hour postprandial glucose incremental area under the curve (IAUC), calculated from blood samples taken 5 min prior to meal, 0, 15, 30, 45, 60, 90 and 120 min after the start of the test meal.
Time Frame: 2 hours
Measure: Mean (Standard Error); unit: mmol*min/L
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
mmol*min/L | 124 (16) | 106 (16)
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 0.087, t-test, 2 sided

2. Secondary Outcome: 2-hour Postprandial Insulin Incremental Area Under the Curve (IAUC)
Description: 2-hour postprandial insulin incremental area under the curve (IAUC) calculated from blood samples taken 5 min prior to meal, 0, 15, 30, 45, 60, 90 and 120 min after the start of the test meal.
Time Frame: 2 hours
Measure: Mean (Standard Error); unit: pmol*h/L
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
pmol*h/L | 245 (24) | 189 (21)
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 0.020, t-test, 2 sided

3. Secondary Outcome: Abdominal Bloating
Description: The occurrence of abdominal bloating (none, mild, moderate or severe) daily before breakfast during the three days of each pre-feeding period and before consuming the test meal on day 4.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
Participants | 8 | 8
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 1.00, Fisher Exact

4. Secondary Outcome: Belching
Description: The occurrence of belching (none, mild, moderate or severe) daily before breakfast during the three days of each pre-feeding period and before consuming the test meal on day 4.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
Participants | 9 | 10
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 0.70, Fisher Exact

5. Secondary Outcome: Nausea
Description: The occurrence of nausea (none, mild, moderate or severe) daily before breakfast during the three days of each pre-feeding period and before consuming the test meal on day 4.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
Participants | 8 | 9
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 0.71, Fisher Exact

6. Secondary Outcome: Diarrhea
Description: The occurrence of diarrhea (none, mild, moderate or severe) daily before breakfast during the three days of each pre-feeding period and before consuming the test meal on day 4.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
Participants | 6 | 7
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 0.71, Fisher Exact

7. Secondary Outcome: Flatulence
Description: The occurrence of flatulence (none, mild, moderate or severe) daily before breakfast during the three days of each pre-feeding period and before consuming the test meal on day 4.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
Participants | 11 | 12
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 0.67, Fisher Exact

8. Secondary Outcome: Satiety Scores
Description: Satiety is the mean of 4 measures, hunger (H), fullness (F), desire to eat (D) and prospective consumption (how much do you think you can eat) (P) each measured using visual analogue scales (VAS) at intervals over the postprandial period. A VAS is a 100mm line anchored at the right end with phrase indicating a high in tensity of the feeling (eg. as hungry as I have ever felt) and at the left other end with a phrase indicating a low intensity of feeling (eg. not hungry at all). For each measure the minimum score is 0 and the maximum score is 100, as measured in mm from the left end. Higher scores mean more hungry, less full, more desire to eat and high prospective consumption (can eat a large amount). The mean score is calculated as (H - F + D + P)/4.
Time Frame: 2 hours
Measure: Mean (Standard Error); unit: mm
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
mm | 79 (9) | 70 (8)
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 0.11, t-test, 2 sided

9. Post Hoc Outcome: 0-90min Incremental Area Under the Glucose Curve
Description: Incremental area under the curve from 0 to 90 min calculated from blood samples taken 5 min prior to meal, 0, 15, 30, 45, 60 and 90 min after the start of the test meal.
Time Frame: 90 min
Measure: Mean (Standard Error); unit: mmol*min/L
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
mmol*min/L | 108 (13) | 87 (12)
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 0.023, t-test, 2 sided

10. Post Hoc Outcome: 0-90min Incremental Area Under the Insulin Curve
Description: as for outcome 9
Time Frame: 90 min
Measure: Mean (Standard Error); unit: pmol*h/L
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
pmol*h/L | 216 (21) | 162 (18)
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 0.014, t-test, 2 sided

11. Post Hoc Outcome: Glucose Peak Rise
Description: Difference between fasting and maximum glucose concentration during the test
Time Frame: 2 hours
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Control Cookie | Fibersym Cookie
Number analyzed (Participants) | 15 | 15
mmol/L | 2.20 (0.24) | 1.72 (0.23)
Statistical Analysis 1: Comparison: Control Cookie vs Fibersym Cookie; Test type: Superiority; p = 0.040, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Control Cookie | Fibersym Cookie
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 1/16 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Cookie (N=16) | Fibersym Cookie (N=15)
Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Deemed to be of moderate severity and not related to the investigational product by the qualified investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT04820322/Prot_SAP_000.pdf